CLINICAL TRIAL: NCT06452732
Title: Using Multiparametric Flow Cytometry to Detect Peripheral Blood and Bone Marrow Leukaemia Stem Cells for Relapse Prediction in Pediatric Acute Myeloid Leukaemia: a Prospective Study
Brief Title: Using Multiparametric Flow Cytometry to Detect Peripheral Blood and Bone Marrow Leukaemia Stem Cells for Relapse Prediction in P-AML
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Chang Yingjun, Chief Physician, Peking University People's Hospital
Other Study IDs: PekingUPH Chang Ying-Jun
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRD monitoring
  Interventions: Other: MFC for the determination of leukemia stem cell

INTERVENTIONS:
Other: MFC for the determination of leukemia stem cell — MFC for the determination of leukemia stem cell

SUMMARY:
Leukaemia is a major disease that seriously endangers human health, the long-term survival rate of acute myeloid leukaemia receiving conventional chemotherapy is only 10% to 45%, haematological relapse is the main cause of treatment failure in acute myeloid leukaemia, reducing the relapse rate is the key to improving the efficacy of acute leukaemia, biomarker-guided preemptive therapy is an effective way to reduce the recurrence of leukaemia, existing markers to predict the recurrence has a high false Existing markers have high false-negative and false-positive rates for predicting relapse, and improving the accuracy of leukaemia relapse prediction is a major clinical problem that needs to be solved urgently. The group has found that circulating leukaemia stem cells remaining after chemotherapy are the key to relapse, therefore, we propose to conduct a multicentre prospective clinical study on the prediction of acute leukaemia relapse by circulating leukaemia stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnoses candidates with acute myeloid leukemia.
* Lower than or equal to 18 years-old;
* Subjects are able to provide written informed consent.

Exclusion Criteria:

* Subjects who cannot comply with the study;
* Subjects with severe cardiac disease (ejection fraction<50% ), liver disease (total bilirubin >34umol/L, ALT and AST>1.5×upper limit normal) or kidney disease (Serum creatinine>130umol/L).
* Subjects with severe infection.
* Subjects with other conditions that cannot receive chemotherapy or transplantation.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study was an exploratory study in search of new biomarkers, based on the previous literature, the recurrence rates of pre-transplant MRD (+) and MRD (-) in pediatric AML were 41% and 23.8% respectively (Br J Haematol.2024;204:585-594), with the ratio of patients in the two groups being 1:1.The calculation was done using PASS 15.0 assuming a two-sided test of α=0.05 and a test efficacy of = 1-β=80%, with the number of people needed being 226, taking into account a 20% censoring rate, the final total sample size was 283 patients.
Sampling Method: Probability Sample
Enrollment: 283 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary end point was cumulative incidences of relapse (CIR) | 2 years
  Relapse was defined by the morphological evidence of disease in the peripheral blood, BM or extramedullary sites. Time to relapse was defined from the date of diagnosis to the date of disease recurrence. Patients exhibiting minimal residual disease were not classified as having relapsed.

SECONDARY OUTCOMES:
Leukemia free survival (LFS) | 2 years
  Leukimia-free survival was defined as days from diagnosis to disease progression after transplantation.
Overall survival (OS) | 2 years
  Overall survival referred to patients who survived until the final follow-up time point.
Non-relapse mortality (NRM) | 2 years
  Non-relapse mortality was defined as all causes of death other than those related directly to malignant disease itself, occurring at any time after CR.
Transplant related mortality (TRM) | 2 years
  Transplant-related mortality was defined as all causes of death other than those related directly to malignant disease itself, occurring at any time after transplantation.
Acute GVHD | 2 years
  Acute GVHD was defined and graded from 0 to IV based on the pattern and severity of organ involvement[Sullivan KM. Graft-versus-host-disease. In: Thomas ED, Blume KG, Forman SJ (eds). Hematopoietic Cell Transplantation. 2nd edn. Blackwell Science: Boston, MA, USA, 1999, pp 515-536.]; grades III-IV aGVHD manifest as serious clinical features on the skin, liver and/or gut.
Chronic GVHD | 2 years
  Chronic GVHD was defined and graded according to the National Institute of Health criteria:[Biol Blood Marrow Transplant,2005,11: 945] that is, mild cGVHD reflects the involvement of no more than 1 or 2 organs/sites (except for lung) with a maximum score of 1; moderate cGVHD involves at least 1 organ/site with a score of 2 or ≥3 organs/sites with a score of 1 (or lung score 1); and severe cGVHD is diagnosed when a score of 3 is given to any organ (or lung score 2). The diagnosis is mainly based on clinical manifestations.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - People's Hospital of Peking University, Beijing, Beijing Municipality